CLINICAL TRIAL: NCT01822080
Title: A Multicenter Study to Investigate the Efficacy and Safety of Daily Oral Administration of 2 mg Dienogest Tablets (Visanne/SH T00660AA) for the Treatment of Endometriosis in Chinese Patients: a Double-blind, Randomized, Placebo-controlled, Parallel Group Phase Over 24 Weeks Followed by an Open-label, Single-group Follow up Over 28 Weeks
Brief Title: Phase 3 Study of Dienogest for the Treatment of Endometriosis in Chinese Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13390
Record Dates: First submitted 2013-03-11; First posted 2013-04-02 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2015-11

CONDITIONS: Endometriosis
Keywords: Endometriosis; Efficacy; Safety; Dienogest
MeSH Terms: conditions — Endometriosis | interventions — dienogest

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dienogest (Experimental): 50% of the participants will be randomized to this arm and will receive 2 mg dienogest (DNG) once daily by mouth from 0-52 weeks
  Interventions: Drug: Dienogest (Visanne, BAY86-5258)
- Placebo (Placebo Comparator): 50% of the participants will be randomized to this arm and will receive placebo once daily by mouth from 0-24 weeks then switch to 2 mg dienogest (DNG) once daily by mouth from 25-52 weeks
  Interventions: Drug: Dienogest (Visanne, BAY86-5258); Drug: Placebo

INTERVENTIONS:
Drug: Dienogest (Visanne, BAY86-5258) — 2 mg dienogest (DNG) once daily by mouth
Drug: Placebo — Matching placebo once daily by mouth
  Arms: Placebo

SUMMARY:
This study is aimed to evaluate efficacy and safety of dienogest 2 mg oral tablets in the treatment of endometriosis.

There will be 2 study phases: a double-blind, randomized, placebo-controlled, parallel-group phase over 24 weeks, and an open-label extension phase with 2 mg DNG daily p.o. over 28 weeks for all subjects who completed the double-blind phase, irrespective of their treatment assignment in the first study phase.

ELIGIBILITY:
Inclusion Criteria:

* Women between 18 and 45 years of age, inclusive
* Women with endometriosis confirmed by laparoscopy or laparotomy within ten years but no later than 2 weeks before the Screening Visit
* A score of at least 30 on a 100 mm visual analog scale (VAS) for endometriosis-associated pelvic pain at Screening Visit and Baseline Visit
* Good general health (except for findings related to endometriosis, with or without infertility), as evidenced by medical history and complete physical and gynecological examination
* Willingness to use a barrier method of contraception is required

Exclusion Criteria:

* Pregnancy or lactation (less than three months since delivery, abortion, or lactation before start of treatment)
* Wish for pregnancy within intended treatment period
* Before menarche or after menopause
* Amenorrhea (more than three consecutive months in the six months before screening)
* Undiagnosed abnormal genital bleeding
* Previous/use of hormonal agents
* Any disease or condition that may worsen under hormonal treatment
* Signs and/or symptoms of therapy-resistant endometriosis despite more than one prior attempt at drug treatment or surgical therapy
* Need for primary surgical treatment of endometriosis
* Regular use of pain medication due to other underlying diseases
* Contra-indication for the supportive analgesic medication (ibuprofen)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 250 (Actual)
Dates: Start 2013-03; Primary Completion 2015-04 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change of endometriosis associated pelvic pain (EAPP) measured by visual analog scale (VAS) from baseline to 24 weeks | 24 weeks after baseline

SECONDARY OUTCOMES:
Percentage of treatment responders | At 24 weeks
Score on B&B (Biberoglu and Behrman severity profile for symptoms and findings) | 24 weeks after baseline
Quality of life assessed by patient questionnaire | Up to 24 weeks
Number of participants with adverse events as a measure of safety and tolerability | Up to 52 weeks
Vaginal bleeding intensity recorded by patient diary and measured on a 5-point scale (none, spotting, light, normal, heavy) | Up to 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (14):
- China (14):
  - Guangzhou, Guangdong
  - Shijiazhuang, Hebei
  - Wuhan, Hubei
  - Hengyang, Hunan
  - Changchun, Jilin
  - Dalian, Liaoning
  - Shenyang, Liaoning
  - Xi'an, Shaanxi
  - Chengdu, Sichuan
  - Hangzhou, Zhejiang
  - Beijing
  - Chongqing
  - Kunming
  - Shanghai

REFERENCES:
- [Derived] Yu Q, Zhang S, Li H, Wang P, Zvolanek M, Ren X, Dong L, Lang J. Dienogest for Treatment of Endometriosis in Women: A 28-Week, Open-Label, Extension Study. J Womens Health (Larchmt). 2019 Feb;28(2):170-177. doi: 10.1089/jwh.2018.7084. Epub 2018 Nov 21. PMID 30461337